CLINICAL TRIAL: NCT07239466
Title: A Single-Arm, Single-Center Study of Exploring the β-hydroxybutyrate Supplementation and Short-Course Radiotherapy Followed by Immunotherapy Combined With CAPEOX Neoadjuvant Therapy in Locally Advanced Rectal Cancer
Brief Title: A Pilot Study Evaluating β-hydroxybutyrate Supplementation Concomitant to Short-Course Radiotherapy Followed by Immunotherapy Combined With CAPEOX Neoadjuvant Therapy in Patients With Locally Advanced Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tao Zhang (Other)
Responsible Party: Sponsor-Investigator, Tao Zhang, MD, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Union-BHB
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Rectal Cancer; Radiotherapy; Immunotherapy; Chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Radiotherapy (SCRT): Total dose 25 Gy delivered in 5 fractions (5 Gy per fraction, once daily over 5 consecutive days).
  β-hydroxybutyrate: Oral β-hydroxybutyrate supplement (5g/day, starting from the day of first radiotherapy, lasting for 2 weeks).
  Immunotherapy (PD-1 monoclonal antibody): 200 mg via intravenous infusion every 3 weeks (q3w) for 2 cycles, initiated 1 week after radiotherapy completion.
  Chemotherapy (CAPEOX regimen): Oxaliplatin: 130 mg/m² IV infusion over 120 minutes on Day 1. Capecitabine: 1000 mg/m² orally twice daily (morning and evening, 30 minutes after meals) on Days 1-14. Cycle duration: 3 weeks per cycle; total of 2 cycles during the neoadjuvant phase.
  Interventions: Radiation: Short-course radiotherapy; Drug: Capecitabine; Drug: Oxaliplatin; Procedure: TME surgery; Dietary Supplement: β-hydroxybutyrate

INTERVENTIONS:
Radiation: Short-course radiotherapy — Eligible subjects will receive short-course radiotherapy (SCRT). One week after the end of treatment, subjects continued to receive neoadjuvant chemotherapy.
Drug: Capecitabine — 1000mg/m2, bid, po, d1-14,q3w
Drug: Oxaliplatin — 130mg/m2, ivgtt, d1,q3w
Procedure: TME surgery — The surgery was performed 1 week after the end of neoadjuvant therapy.
Dietary Supplement: β-hydroxybutyrate — Oral β-hydroxybutyrate supplement (5g/day, starting from the day of first radiotherapy, lasting for 2 weeks).

SUMMARY:
This study is a prospective phase II clinical trial aimed at exploring the potential benefits of supplementing β-hydroxybutyrate with existing short course radiotherapy sequential immunotherapy and CAPEOX therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their family members agree to participate in the study and sign the informed consent form;
2. Age 18-75 years, male or female;
3. Histologically confirmed Locally Advanced rectal adenocarcinoma;
4. inferior margin ≤ 10 cm from the anal verge;
5. ECOG performance status score is 0-1;
6. Untreated with anti-tumor therapy for rectal cancer, including radiotherapy, chemotherapy, surgery, etc;
7. There was no operative contraindication;
8. Laboratory tests were required to meet the following requirements: white blood cell (WBC) ≥ 4×109/L; Absolute neutrophil count (ANC) ≥ 1.5×109/L; Platelet count ≥ 100×109/L; Hemoglobin ≥90 g/L; Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN); Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; Serum creatinine ≤1.5 times the upper limit of normal value or creatinine clearance rate ≥50 mL/min; International normalized ratio (INR) ≤ 1.5 × ULN; Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;
9. Urinary protein < 2+ or 24-hour urinary protein excretion < 1 g at baseline.

Exclusion Criteria:

1. Patients with non-pMMR LARC；
2. Subjects who have previously received any form of immunotherapy, including but not limited to immune checkpoint inhibitors, immune checkpoint agonists, immune cell therapy, or any other treatment targeting tumor immunomodulatory mechanisms;
3. Presence of any concurrent disease, condition (including laboratory abnormality), history of substance abuse, or current evidence thereof, which, in the judgment of the Investigator, may compromise subject safety, interfere with the process of obtaining informed consent, affect subject compliance, or confound the safety assessment of the investigational product(s).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) rate | an expected average of 12 months
  Defined as pathological complete response (pCR) + Clinical complete response (cCR)

SECONDARY OUTCOMES:
3-year disease-Free Survival | an expected average of 3 years
  The time from the first day of disease free (operation date) to local or distant recurrence, or the death event caused by any reason, whichever occurs first
Overall Survival | an expected average of 5 years
  The time from the date of randomization to the death caused by any cause
Adverse events (AEs) were graded according to the NCI CTCAE version 5·0 | an expected average of 1.5 years
  Adverse events and surgical safety

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Lin, Principal Investigator — Huazhong University of Science and Technology Tongji Medical College Union Hospital
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided